CLINICAL TRIAL: NCT04284943
Title: A Randomized Controlled Trial Comparing Billroth II Reconstruction Versus Conventional Roux-en-Y Reconstruction Versus Long Limb Roux-en-Y Reconstruction for Glycemic Control in Patients With Concurrent Type 2 Diabetes and Gastric Cancer
Brief Title: Surgical TreAtment for Obesity Related Disease and Onco-Metabolic Surgery
Acronym: STARDOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); The First Hospital of Jilin University (Other); Shanghai Jiao Tong University School of Medicine (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Korea University Ansan Hospital (Other)
Responsible Party: Principal Investigator, Sungsoo Park, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STARDOM
Record Dates: First submitted 2020-02-23; First posted 2020-02-26 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Gastric Cancer; Diabetes Mellitus, Type 2
Keywords: Gastric Cancer; Diabetes Mellitus, Type 2; Subtotal Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Long limb Roux-en-Y reconstruction (Active Comparator): Long limb Roux-en-Y reconstruction method follows subtotal gastrectomy for gastric cancer.
  Interventions: Procedure: Long limb Roux-en-Y reconstruction after subtotal gastrectomy
- Conventional Roux-en-Y reconstruction (Active Comparator): Conventional Roux-en-Y reconstruction method follows subtotal gastrectomy for gastric cancer.
  Interventions: Procedure: Conventional Roux-en-Y reconstruction after subtotal gastrectomy
- Billroth II reconstruction (Active Comparator): Billroth II reconstruction method follows subtotal gastrectomy for gastric cancer
  Interventions: Procedure: Billroth II reconstruction after subtotal gastrectomy

INTERVENTIONS:
Procedure: Long limb Roux-en-Y reconstruction after subtotal gastrectomy — The jejunum will be divided approximately 150 cm distal to the ligament of Treitz (Length of biliopancreatic limb). The gastrojejunostomy will be performed by end-to-end anastomosis and an anastomosis of the proximal end of the jejunum to the distal jejunum will be created approximately 50 cm distal from the gastrojejunal anastomosis (Length of Roux-en-Y limb).
  Arms: Long limb Roux-en-Y reconstruction
Procedure: Conventional Roux-en-Y reconstruction after subtotal gastrectomy — The jejunum will be divided approximately 20 cm distal to the ligament of Treitz (Length of biliopancreatic limb). The gastrojejunostomy will be performed by end-to-end anastomosis and an anastomosis of the proximal end of the jejunum to the distal jejunum will be created approximately 30-45 cm distal from the gastrojejunal anastomosis (Length of Roux-en-Y limb).
  Arms: Conventional Roux-en-Y reconstruction
Procedure: Billroth II reconstruction after subtotal gastrectomy — The duodenum will be transected approximately 2 cm distal to the pylorus and anastomosis will be performed between the gastric remnant and a loop of jejunum chosen approximately 20 cm distal to the ligament of Treitz (Length of afferent loop)
  Arms: Billroth II reconstruction

SUMMARY:
This is a prospective, multi-center, randomized controlled trial to compare Billroth II reconstruction versus conventional Roux-en-Y reconstruction versus long limb Roux-en-Y reconstruction for glycemic control in patients with concurrent type 2 diabetes and gastric cancer.

DETAILED DESCRIPTION:
Billroth I, Billroth II, or Roux-en-Y procedure follows gastrectomy to reconstruct the gastrointestinal tract. Billroth I procedure restores the normal configuration of the gastrointestinal tract and Billroth II and Roux-en-Y procedure involve the creation of duodenal switch which is thought to be responsible for metabolic effects by altering enteric hormones. Accordingly, several retrospective studies reported that Billroth I reconstruction has less effect on diabetes compared to Billroth II and Roux-en-Y reconstruction. While little is known about different effects of Billroth II and Roux-en-Y procedure, a study retrospectively show that Roux-en-Y procedure has significantly higher rate of T2DM remission than Billroth II procedure. Investigators conduct a randomized controlled trial to control possible confounders arising from diverse metabolic effects of cancer and minimize differences in treatment regimen among patients.

ELIGIBILITY:
Inclusion Criteria:

* Distal gastric adenocarcinoma diagnosed pathologically under preoperative endoscopic biopsy, and clinical stage I-II
* Body mass index ≥ 23 kg/m2
* Type 2 diabetes and HbA1c ≥ 6.5%

Exclusion Criteria:

* Insulin usage for glycemic control at the time of screening evaluation
* Prior gastrointestinal surgery including splenectomy, hepatobiliary and pancreatic surgery (except hemorrhoidectomy, herniorrhaphy, and appendectomy)
* Abdominal, thoracic, pelvic and/or obstetric-gynecologic surgery within 3 months
* Cardiovascular conditions including significant known CAD, uncompensated congestive heart failure, history of stroke, or uncontrolled hypertension. Subjects with CAD that have been successfully treated with CABG or PCI, and have no evidence of active ischemia are eligible
* Kidney disease including renovascular hypertension, renal artery stenosis, or end-stage renal disease
* Chronic liver disease including liver cirrhosis, alpha-1 antitrypsin deficiency
* Gastrointestinal disorders including inflammatory bowel disease (Crohn's disease or ulcerative colitis) or any malabsorptive disorders
* Psychiatric disorders including dementia, active psychosis, history of suicide attempts, alcohol or drug abuse within 12 months
* Severe pulmonary disease defined as FEV1 <50% of predicted value
* Anemia defined as hemoglobin less than 8 in females and 10 in males
* Malignancy within 5 years (except squamous cell and basal cell cancer of the skin). Subjects diagnosed with early or stage I cancer than have been successfully treated are eligible per investigator discretion
* Frail elderly (Rockwood Clinical Frailty Scale ≥5)
* Any condition or major illness that, in the investigator's judgement, places the subject at undue risk by participating in the study
* Unable to understand the risks, realistic benefits and compliance requirements of each program
* Use of investigational therapy or participation in any other clinical trial within 3 months
* Geographic inaccessibility
* Pregnancy

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The success rate of biochemical improvement of diabetes as measured by HbA1c < 6.5% | 12 months
  The proportion of subjects with HbA1c < 6.5% without diabetes medications

SECONDARY OUTCOMES:
Time to first occurence of glycated hemoglobin < 6.5% (or 6.0%) | Every visit date, assessed up to 12, 24, and 36 months
  The number of days from randomization to the visit date when HgA1c is first observed to be < 6.5% (or 6.0%) post-randomization
Success rate of biochemical resolution of diabetes | 12 months, 24 months, 36 months
  Success rate of biochemical improvement of diabetes at 12, 24, 36 months as measured by HbA1c ≤ 6% (with or without diabetes medication)
Success rate of biochemical improvement of diabetes | 12 months, 24 months, 36 months
  Success rate of biochemical improvement of diabetes at 12, 24, 36 months as measured by HbA1c <6.5% (with or without diabetes medication)
Change in glycated hemoglobin from baseline | 12 months, 24 months, 36 months
  percent change
Change in fasting plasma glucose level from baseline | 12 months, 24 months, 36 months
  percent change
Change in total cholesterol | 12 months, 24 months, 36 months
  Percent change in total cholesterol at 12 months, 24 months, 36 months
Change in triglyceride | 12 months, 24 months, 36 months
  Percent change in triglyceride at 12 months, 24 months, 36 months
Change in High-density Lipoprotein (HDL) | 12 months, 24 months, 36 months
  Percent change in high-density lipoprotein (HDL) at 12 months, 24 months, 36 months
Change in Low-density Lipoprotein (LDL) | 12 months, 24 months, 36 months
  Percent change in Low-density Lipoprotein (LDL) at 12 months, 24 months, 36 months
Use of diabetes medication | 12 months, 24 months, 36 months
  number of diabetes medication at 12 months, 24 months, 36 months
Patients with hypertension and/or requiring antihypertensive therapy | 12 months, 24 months, 36 months
  number and percentage
Patients with dyslipidemia and/or requiring cholesterol lowering medications | 12 months, 24 months, 36 months
  number and percentage
Mean and change in weight and BMI from baseline | 12 months, 24 months, 36 months
  mean and percent change
Mean and change in waist, hip, and thigh circumference from baseline | 12 months, 24 months, 36 months
  mean and percent change
Change in SF-36 scores of questionnaire from baseline | 12 months, 24 months, 36 months
  The MOS 36-Item Short-Form Health Survey
Change in High-sensitivity C-reactive Protein (Hs-CRP) | 12 months, 24 months, 36 months
  percent change in high-sensitivity C-reactive protein (hs-CRP)
Change in Systolic Blood Pressure (SBP) | 12 months, 24 months, 36 months
  Change in Systolic Blood Pressure (SBP) at 12 months, 24 months, 36 months
The Side Effects and /or Complications of each surgical procedure | 12 months, 24 months, 36 months
  number of the Side Effects and /or Complications of each surgical procedure
The success rate of biochemical improvement of diabetes as measured by HbA1c < 6.5% | 24 months, 36 months
  The proportion of subjects with HbA1c < 6.5% without diabetes medications

CONTACTS AND LOCATIONS:
Overall Officials: Sungsoo Park, MD, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No